CLINICAL TRIAL: NCT01190826
Title: Single-Center, Randomized, Double-Blind, Placebo-Controlled, Three-Way Crossover Study to Evaluate the Safety, Tolerability and Clinical Activity of a Single Dose of ASM-024 Administered by Inhalation to Subjects With Stable Moderate Asthma
Brief Title: Safety, Tolerability and Clinical Activity of ASM-024 in Stable Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asmacure Ltée (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ASM-024/II/STA-02
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: Stable moderate asthma
MeSH Terms: conditions — Asthma | interventions — ASM-024

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASM-024 10 mg (Experimental): ASM-024 administered once by inhalation at a target dose of 10 mg
  Interventions: Drug: ASM-024
- ASM-024 100 mg (Experimental): ASM-024 administered once at a target dose of 100 mg
  Interventions: Drug: ASM-024 100 mg
- Placebo (Placebo Comparator): Placebo administered once by inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASM-024 — Target dose of 10 mg ASM-024 administered once by inhalation
  Arms: ASM-024 10 mg
Drug: ASM-024 100 mg — Target dose of 100 mg ASM-024 administered once by inhalation
  Arms: ASM-024 100 mg
Drug: Placebo — Placebo administered once by inhalation
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and clinical activity of ASM-024 in stable moderate asthma.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent.
* Male or female subjects, ≥ 18 years and ≤ 55 years of age
* Diagnosis of moderate asthma and on regular inhaled corticosteroids with or without short or long-acting Beta-2-agonists
* FEV1 ≥ 55 % predicted in the absence of medications for asthma
* Female subjects of childbearing potential must have a negative pregnancy test (serum beta-human chorionic gonadotropin (b-HCG)) at Screening, and a negative pregnancy test immediately before the administration of the study drug for each of Periods 1, 2 and 3. Sexually active females with non-sterile partner must be willing to use adequate contraception.
* Male subjects must be willing to use a condom with a spermicide for the duration of their participation in the study, plus an additional 30 days following study drug administration and ensure that their partner is using a highly effective method of birth control such as combined oral contraceptives, implants, injectables or an intra-uterine device (IUD). Male subjects must ensure that their female partner is willing to use adequate contraception.
* Demonstration of an increase in FEV1 by ≥ 10 % predicted between spirometry performed before and 10-20 minutes after the administration of 2 puffs of 100 micrograms of salbutamol at Screening.

Exclusion Criteria:

* Clinically significant conditions or illnesses other than moderate asthma or systemic diseases
* Pregnant or nursing women or women intending to conceive during the course of the study or have a positive serum pregnancy test at Screening or a positive urine pregnancy test during the study.
* Women of childbearing potential (unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years) not using a highly effective method of birth control.
* Non-surgically sterile males and males with partners of childbearing potential not willing to use a condom with spermicide for the duration of their participation in the study plus an additional 30 days following study drug administration and to ensure that their partner is using a highly effective method of birth control such as combined oral contraceptives, implants, injectables or an IUD.
* Respiratory tract infections or worsening of asthma or changes in asthma medications within 6 weeks before Screening/Baseline.
* Current cigarette smokers or former smokers with a smoking history of greater than 10 pack years or who stopped smoking within 12 months preceding enrolment in the study.
* Positive urine cotinine test at Screening.
* History of illicit drug use or alcohol abuse within 12 months before Screening.
* Positive test for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV) at Screening.
* Any medication that are known to prolong QT / QTc interval.
* Any of the following concomitant medications preceding the administration of salbutamol during Screening and preceding the administration of the study drug:

  * Oral or i.v. corticosteroids within 1 month;
  * Inhaled or intranasal corticosteroids within 48 hours;
  * Long acting Beta-2-agonists within 24 hours;
  * Short acting Beta-2-agonists within 8 hours;
  * Anticholinergic aerosols within 24 hours; and
  * Theophylline-containing products within 48 hours.
* Use of NSAIDs within 7 days preceding the administration of salbutamol during Screening and throughout the study.
* Use of antihistaminic drugs within 3 days preceding the administration of salbutamol during Screening.
* Use of an investigational product or participation in a clinical trial using an investigational product within 30 days before dosing or within 90 days in the case of long-acting products (ex.: Depo-medrol) or biologics with a long-acting half-life (ex.: monoclonal antibodies).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Peak change in FEV1 following inhalation of ASM-024 | Over a period of 6 hours following administration

SECONDARY OUTCOMES:
FEV1 AUC following inhalation of ASM-024 | Over 6 hours following administration

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, B. Pharm. MD, Principal Investigator — Anapharm
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Anapharm, Montreal, Quebec
  - Centre de Recherche Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec